CLINICAL TRIAL: NCT06630195
Title: Nature and Frequency of Genetic Abnormalities and Associated Phenotypes in a Cohort of Adults With Intellectual Disability
Acronym: HiNDIA
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231767
Record Dates: First submitted 2024-09-09; First posted 2024-10-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-09

CONDITIONS: Intellectual Disabilities
Keywords: Phenotypes; intellectual disabilities; genetic abnormalities
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Intellectual disability (ID) is characterized by having an intelligence quotient (IQ) below 70 and substantial limitations in adaptive functioning across different domains, with the condition manifesting before the age of 18. Historically, it was noted that 25% of ID cases were attributed to acquired causes such as perinatal anoxia or infections, another 25% were linked to genetic factors, and the remaining 50% had an 'undetermined' cause. However, with advancements in genetic diagnosis, the proportion of cases with unknown causes is gradually diminishing, giving way to a greater understanding of genetic etiologies. The rarity of each of these causes of ID and the lack of specificity of most of the syndromes mean that it is often difficult to make an aetiological diagnosis. The objective of this study is to describe the nature and frequency of genetic abnomalties identified in adult patients with intellectual disability.

This is a descriptive, retrospective and prospective study that aim to include 1000 patients across 10 centres aged over 20 years old on consultation between 2016 to 2025 who have been informed (where applicable, the guardian), who have not oppose to participate and who meet the inclusion and non-inclusion criteria. Each centre will include and increment a patient identification number for pseudonymisation of reports. A name correspondence table will be maintained by each center to establish a link between the research identifier and the participant's identity. Each table will be stored on each centre's secure server. The anonymized reports will be transmitted to the coordinating team through the secure Dispose platform, which will transfer all the participants' data to a REDCap APHP database. Descriptive statistic will be performed to count the number of patients with the same genetic syndrome. The age of onset of comorbidities and the proportion of each complication by syndromes will be calculated for all patient, including the means and median.

DETAILED DESCRIPTION:
Intellectual disability (ID) is defined by the combination of an intelligence quotient (IQ) of less than 70 and significant limitations in adaptive functioning in various areas, with onset before the age of 18. Although common (2% of the population), ID is an extremely heterogeneous condition in terms of severity, associated additional disabilities and aetiologies. Until recently, it was reported that 25% of IDs had an acquired cause (perinatal anoxia, infection, etc.), 25% a genetic cause, and 50% an 'undetermined' cause; advances in genetic diagnosis are gradually reducing the latter proportion in favour of genetic aetiologies. The rarity of each of the genetic causes of ID and the lack of specificity of most of the syndromes mean that it is often difficult to make an aetiological diagnosis.

This is a descriptive, retrospective and prospective study that aim to include 1000 patients across 10 centres aged over 20 years old on consultation between 2016 to 2025 who have been informed (where applicable, the guardian), who have not oppose to participate and who meet the inclusion and non-inclusion criteria. The first stage of the study will be the selection of patients' medical records by the participating centres. Patients aged over 20 with a proven intellectual disability who have been seen for consultations since 2016 will be identified on the basis of their electronic and/or paper medical records (retrospetive). Selection of the file includes a check of the elements present and missing from the file, using a clinical data collection grid and genetic results. If the data is available, the patient will then be selected. Once the files have been selected, the patient or, where appropriate, the guardian (if the patient is under guardianship) will be informed individually of the study and asked for their non opposition. For the prospective arm, patients over the age of 20 with a proven intellectual disability who are seen for routine care in the participating centres will be included. Each centre will increment a patient identification number for pseudonymisation of reports. A name correspondence table will be maintained by each center to establish a link between the research identifier and the participant's identity. Each table will be stored on each centre's secure server. The anonymized reports will be transmitted to the coordinating team through the secure Dispose platform, which will transfer all the participants' data to a REDCap APHP database.

Descriptive statistic will be performed to count the number of patients with the same genetic syndrome. The age of onset of comorbidities and the percentage of each complication per syndrome will be calculated for all patients, including the means and median.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 20 years of age with a proven intellectual disability,
2. Patient seen in consultation between 2016 and 2025
3. No objection from the patient or, where applicable, the guardian

Exclusion Criteria:

1. Medical file not available
2. Opposition from the patient or, where applicable, the guardian.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 20 years of age with a proven intellectual disability, seen in consultation between 2016 and 2025
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
List and frequency of genetic anomalies identified in adults with an intellectual disability | Through study time period (24 months)

SECONDARY OUTCOMES:
Describe the clinical phenotype in adulthood corresponding to the genetic anomalies identified, with particular attention to adults over 45 years of age | Through study time period (24 months)
Describe the co-morbidities and complications of genetic syndromes over time | Through study time period (24 months)
Evaluate the frequency of genetic diagnosis in adults with ID | Through study time period (24 months)

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.